CLINICAL TRIAL: NCT07137442
Title: Distinguishing Tics and Functional Tics Using Clinical Neurophysiological Techniques
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002309; 002309-N
Record Dates: First submitted 2025-08-19; First posted 2025-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-12

CONDITIONS: Tics; Functional Tics
Keywords: Tics; Functional tics; EEG; Blink Reflex; Pre-pulse inhibition
MeSH Terms: conditions — Tics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Functional Tics: Individuals with tics as the phenomenology of functional movement disorder. The functional tics convey a condition of tics in which the primary pathophysiological processes are alterations in functioning of brain networks rather than abnormalities of brain structures.
- Healthy controls: Participants without tics or other neurological or active psychiatric disorders.
- Tics: A tic is a sudden, brief and repetitive motor movement or vocalization that is not rhythmic and involves discrete muscle groups.

SUMMARY:
Background:

Tics are involuntary movements and vocalizations. Some tics are organic: They are related to diagnosed disorders. Sometimes tics have other causes, such as problems with how the brain and body send and receive messages. These are called functional tics. It can be difficult to tell the difference between these 2 types of tics. Doctors need to know more so they can make more accurate diagnoses.

Objective:

To learn more about the difference between functional and organic tics.

Eligibility:

Adults aged 18 to 80 years who have a tic that causes involuntary movements. Healthy volunteers with no tics are also needed.

Design:

Participants will have one 4-hour clinic visit. The visit may be done in 1 or 2 days. Participants will refrain from consuming alcohol or caffeine before the visit. They may have a physical exam.

Participants will wear two types of sensors:

Electromyography (EMG): Adhesive disks with sensors will be attached to the skin above some muscles. These disks will record electricity in the muscles as the participant moves.

Electroencephalography (EEG): Sensors will be placed on the participant s scalp. The sensors may be adhered directly, or the participant may wear an electrode cap. The sensors will detect brain waves.

Participants will rest while seated in a chair. Their involuntary tics will be monitored with the EMG and EEG. Then they will be asked to make movements to mimic their tics. Healthy volunteers will also rest; then they will be asked to perform movements that mimic tics.

Participants will have their blink reflex tested. EMG sensors will be placed on the muscles near the eyes. Electrical pulses will be used to stimulate blinking.

Participants will answer questionnaires about their tics and their health....

DETAILED DESCRIPTION:
Study Description:

The purpose of the protocol is to explore the physiological difference between patients with tics and functional tics.

Objectives:

Primary Objective: To determine if there are differences in cortical excitability before tics in patients with tics compared to functional tics.

Secondary Objectives: N.A.

Exploratory Objectives: To determine if there are differences in cortical and subcortical excitability before tics in patients with tics compared to functional tics.

Endpoints:

Primary Endpoint: This is a hypothesis-driven study. The primary outcome measure is the beta power of EEG signal before the tics at

the electrode over the vertex.

Secondary Endpoints: N.A.

Other exploratory outcome measures include EEG signal power across different frequency bands and Bereitschaftspotential at various electrodes with different movements. Blink reflex and pre-pulse inhibition will also be measured in patients with tics and functional tics and healthy controls under different conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Capacity to provide informed consent (self-consent)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-80
* Agreement to adhere to Lifestyle Considerations prior to and during the physiological testing visit.

Inclusion criteria for patients with functional tics or tics

- Diagnosed with functional motor tics or motor tics

Inclusion criteria for healthy controls

- Have no neurological or psychiatric disorders established by history and physical/neurological examination

EXCLUSION CRITERIA:

* Self-reported consumption of >14 alcoholic drinks/week* for a man and >7 alcoholic drinks/week for a woman
* Use of prescription drugs and other illicit drugs that may suppress tics such as dopamine blocking agents and antipsychotics during a certain time period prior to the

neurophysiological testing session.**

* Clinically significant abnormal movements on neurological examination except for tics.
* Contraindications to EEG or EMG procedures, including skin lesions at electrode sites or hypersensitivity to electrode materials.
* History of or current brain tumor, stroke, head trauma with loss of consciousness.
* Epilepsy or seizures in the past 12 months.
* Have a Baclofen pump, or have neurostimulators for pain.
* Pregnant women
* Self-reported current major depression or Beck Depression Inventory II (BDI-II) score >19, Generalized Anxiety Disorder 7-item scale (GAD-7) score > 9, or any major current psychiatric illness.
* Presence of any metal in the eye or skull area such as a brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, metal fragments in the eye.
* Presence of pacemaker, intracardiac lines, implanted pumps or stimulators.
* Unable to comply with the requirements of the study procedures.
* Vocal tics only tested with Modified Rush Video-Based Tic Rating Scale.
* Low Premonitory Urge for Tics Scale (PUTS) score < 9 (maximum 36) with low willingness for tics (patient groups only, not applicable in healthy volunteers).

  * Note: 1 standard alcoholic drink is 0.6 ounce (14 grams) of pure alcohol.

    * Note: The certain time period depends on different drugs used. Five half-lives will be selected. The drug is considered effectively eliminated from the body after this time period because the concentration of the drug reaches around 3% of the orininal concentration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups with up to 25 subjects in each group. Two groups of patients (18-80 years old) with tics and functional tics, and another group of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2034-08-01 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability as determined by beta power at the vertex | 2 days
  To determine that the cortical excitability excitability before functional tics are different from those before other tics.

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002309-N.html